CLINICAL TRIAL: NCT03825666
Title: Can Simple Perioperative Measures Improve Quality of Recovery Following Ambulatory Laparoscopic Surgery in Females? An Open Prospective Randomised Study, Comparing Nutritional Preoperative Drink and Chewing Gum During Recovery to Standard Care.
Brief Title: Can Simple Perioperative Measures Improve Quality of Recovery Following Ambulatory Laparoscopic Surgery in Females?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, EmmaObrink, Principal Investigator, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Obrink2
Record Dates: First submitted 2019-01-23; First posted 2019-01-31 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Quality of Recovery
Keywords: quality of recovery; PONV; PDNV
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Intervention with drink pre surgery and chewing gum post surgery. No subgroups, combined intervention will be assessed. ProvideXtra® Fresenius Kabi plus standard consumer xylitol chewing gum.
  Interventions: Other: ProvideXtra® Fresenius Kabi
- Control (No Intervention): control group following standard guidelines

INTERVENTIONS:
Other: ProvideXtra® Fresenius Kabi — Improving wellbeeing
  Other Names: standard consumer xylitol chewing gum
  Arms: Active

SUMMARY:
The aim of this study was to assess whether it was possible to improve patients' self-assessed quality of recovery and reduce the level of post-operative nausea and vomiting in female patient undergoing laparoscopic cholecystectomy by simple perioperative measures in the form of a preoperative 200 ml nutritional drink and chewing gum during early recovery.

Patients were randomised to an active group receiving the intervention, and controls provided with standard care only. Patients were followed by questionnaire interviews preoperatively and at 2, 24 and 48 hours after surgery.

DETAILED DESCRIPTION:
Abstract One major goal in modern perioperative anaesthesia care is to facilitate a rapid, yet safe recovery process, with focus on improving time to regained consciousness and subsequent resuming of activities of daily living. Laparoscopic cholecystectomy and gynaecological laparoscopy are a "high volume" procedure commonly performed in young females expecting rapid resumption of health.

The aim of this study was to assess whether it was possible to improve patients' self-assessed quality of recovery and reduce the level of post-operative nausea and vomiting in female patient undergoing laparoscopic cholecystectomy by simple perioperative measures in the form of a preoperative 200 ml nutritional drink and chewing gum during early recovery.

Methods Patients were randomised to an active group receiving the intervention, and controls provided with standard care only. Patients were followed by questionnaire interviews preoperatively and at 2, 24 and 48 hours after surgery. The Quality of Recovery scale (QoR) 15 items and 5 additional questions around gastro-intestinal symptoms were self-assessed by patients at each occasion.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2

Exclusion Criteria:

* ASA 3-4, obese

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Quality of recovery, QoR15, (Quality of Recovery 15) | 48 hours
  Quality of recovery after laparoscopic surgery with a valid questionnaire. 15 questions, max point 150. 0 worse, 10 best score. Mean sum is going to be compared.

IPD SHARING:
Plan to Share IPD: No